CLINICAL TRIAL: NCT05037448
Title: Me & My Wishes: An Efficacy Trial of Long Term Care Residents With Alzheimer's Using Videos to Communicate Care Preferences With Caregivers
Brief Title: Exploring Telehealth to Deliver Me & My Wishes During Coronavirus-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Brown University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gail Towsley, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I00111417
Record Dates: First submitted 2021-08-24; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-03

CONDITIONS: Health Communication

STUDY DESIGN:
Intervention Model Description: The investigators propose to examine the plausibility of delivering Me & My Wishes using a telehealth platform. A convenience sample of five residents, their family members and long term care staff will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth (Other): Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.
  Interventions: Behavioral: Me & My Wishes

INTERVENTIONS:
Behavioral: Me & My Wishes — Me & My Wishes videos communicate residents' preferences via personalized video recorded conversations. Me & My Wishes are videos of nursing home residents talking about their preferences for care, and include four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts.

SUMMARY:
Due to Coronavirus-19, we are exploring the plausibility of delivering the Me & My Wishes intervention via telehealth.

DETAILED DESCRIPTION:
Me & My Wishes are videos of nursing home residents talking about their preferences for care, including four sections: About Me, Preferences for Today, Preferences for Medical Intervention and End of Life, and Afterthoughts. Knowing what residents want is essential to staff's ability to provide quality care and can inform family caregivers decision making especially in later stages of life as the resident's cognition declines-a time when family caregivers often feel unprepared. Persons with mild to moderate dementia can accurately express their everyday and end of life preferences, however, stereotypes persist about the decision making abilities of people with dementia that often prevent their involvement in conversations about care. The investigators propose to explore the feasibility of delivering Me & My Wishes via a telehealth platform.

ELIGIBILITY:
Resident Inclusion Criteria:

* Identified as having Alzheimer's or related dementia
* Mild to moderate cognitive impairment (BIMS = 8-15, (MDS C0500) (nursing home residents only)
* Makes Self Understood = <1 (MDS B0700)/present in medical record
* Understood By Others = <1 (MDS B0800)/present in medical record
* Reside at the facility at least 2 weeks identified as a long-term resident
* Age >65 years
* Speaks English

Family Inclusion Criteria:

* Speaks English
* Willing and able to watch the videos
* Willing to complete short surveys. Being unable to attend care conference to view the video (e.g. due to distance) will not exclude family from participating.

Staff Inclusion Criteria:

* Speaks English
* Willing to watch the videos
* Willing to complete short surveys

Resident Exclusion Criteria:

* Limited communication capacity (e.g. aphasia)
* Comatose
* Cognitively intact
* Severe cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of telehealth-delivered Me & My Wishes | baseline
  ease of use, connecting to internet, communicating with participants. 1-5 scale 1 = strongly disagree, 5 = strongly agree; we also asked what worked well and what could go better
Feasibility of telehealth-delivered Me & My Wishes | 90 days
  ease of use, connecting to internet, communicating with participants. 1-5 scale 1 = strongly disagree, 5 = strongly agree; we also asked what worked well and what could go better

CONTACTS AND LOCATIONS:
Overall Officials: Gail Towsley, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Marquis Forest Grove Post Acute Rehab, Forest Grove, Oregon
  - Marquis Wilsonville Assisted Living, Wilsonville, Oregon
  - Mission at Maple Springs, Brigham City, Utah

IPD SHARING:
Plan to Share IPD: No